CLINICAL TRIAL: NCT03453229
Title: Measurement of FEV1 and Other Physiological Parameters by Connected Devices in Lung Transplanted Patients
Brief Title: Wearable Devices to Assess Physiological Parameters in Lung Transplant Patients
Acronym: EOLE VAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2016GTT1058; 2017-A01908-45 (Other: IDRCB)
Record Dates: First submitted 2018-01-02; First posted 2018-03-05 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Patients Who Received Lung Transplantation (Previous Year)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study will be a prospective non-interventional study involving 15 to 20 lung transplant patients. The patient will do as usual Forced Expiratory Volume (FEV1) measures and some physiological parameters will be automatically recorded through the wearable and wireless sensors. The spirometer will also be connected but only to transmit stored data, not for real time use. The patient and the physician will not have access to the data until the end of the study. The 6 following physiological parameters will be recorded: heart rate, respiratory rate, body temperature, SPO2, motion, and sleep. The study duration for each patient will be 6 months.

The primary endpoint will be the number of FEV1 measures combined with physiological parameters. This primary endpoint has been chosen because it is easy to obtain. The secondary endpoints will be: - physiological parameters associated with a 10% or higher decrease in FEV1, - correlation between variations of physiological parameters and occurrence of a clinical event (defined by presumption of infection or of graft failure), - interval between the first significant modification of each physiological parameter and the onset of an event, - number of recorded values, - patient's satisfaction. In this pilot phase, there is no real time health advice.

DETAILED DESCRIPTION:
Justification of the study: The two main complications responsible for death among lung transplant patients are infection and rejection. In-hospital, 1-year and 5-year mortality is 10%, 20%, and 50%, respectively. The main symptoms are dyspnea, fever, drop in oxygen saturation, drop in pulmonary function tests (FEV1). Investigators hypothesize that surveillance of FEV1 and of several physiologic parameters though connected devices could improve early diagnostic of complications, namely rejection and infection. Surveillance of these patients through connected devices could reduce both mortality and morbidity.

Design of the study: Prospective, observational, monocentric study (Bichat-Hospital, Université Paris 7, France) Main objectives and main endpoint: the main objective is to describe the natural trend of six physiologic parameters (SpO2, heart rate, respiratory rate, cutaneous temperature, physical activity and quality of sleep) and of FEV1 in patients who have benefited from lung transplantation within one year) and to specifically assess the evolution of these parameters a few days before the occurrence of complications. The main criteria of judgment will be mean and standard deviation of these parameters five days before the occurrence of an event, defined by hospitalization for infection and/or graft rejection.

Secondary objectives and secondary endpoints:

The secondary objectives will be:

* To validate metrologic performances of the connected devices.
* To describe the modifications of the physiologic parameters within days before a drop of 10% of FEV1
* To describe the modifications of the physiologic parameters before the occurrence of complications requiring anti-infective and/or anti reject therapies
* To evaluate the interval between modifications of physiologic parameters and the occurrence of infection and/or reject.
* To evaluate the acceptability for the patient and the compliance of connected devices.

The secondary criteria of judgment will be:

* The agreement between physiologic parameters measured through the connected devices and those measured with usual method ("gold standard) during visits in the day-care center
* The mean and standard deviation of the physiologic parameters (including FEV1) recorded for each patient
* The effect of combined physiologic parameters to predict a 10% drop in FEV1, and/or the occurrence of infection and/or the occurrence of graft rejection within 5 days after measurement.
* The interval in days between substantial modifications of physiologic parameters and the occurrence of infection and/or graft rejection.
* The patient's satisfaction measured with a simple questionnaire.

Inclusion criteria

* Adult patients older than 18-years
* Mono or pulmonary transplantation whatever the cause, within the last 12 months
* Inform consent given
* Skill to use connected devices Exclusion criteria
* No exclusion criteria

The devices and the App

Each patient will receive a health kit with the following:

* An App with an electronic formulary allowing the implementation of relevant clinical items: dyspnea, cough, sputum characteristics
* A smartphone
* A connected spirometer
* Wearable devices to record the physiologic parameters.

Duration of the study

Inclusion period: 6 months, Duration of follow-up: 6 months Total duration of the study: 12 months Statistical analysis The distributions of physiologic parameters will be described through mean+/- SD. The comparison of distribution of each physiologic parameter within five days before an event (infection/graft rejection) will allow to define regions in parameter's space associated with an increase in the risk of subsequent events occurrence. For these regions, sensitivity and specificity for predefined thresholds will be calculated. For each event, we will calculate the interval between the entry in a risk region and the occurrence of the event. The standard curve between values recorded through the connected devices and those recorded with the reference measures determined in the hospital will be evaluated with a Bland-Altman representation. The satisfaction questionnaire will be analyzed according to standard methods (distribution of each item, Cronbach alpha coefficient, factorial analyses.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old
* pulmonary transplant less than a year - consantant - mastering the connected tool

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-07-04 (Estimated)

PRIMARY OUTCOMES:
time series of SpO2 (in %) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)

SECONDARY OUTCOMES:
time series of FEV1 (% of theoretical value) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)
time series of Heart rate (in bpm) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)
time series of cutaneous temperature (in °C) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)
time series of respiratory rate (in cycles per minute) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)
time series of physical activity level (measured in a continuous proprietary scale) | 6 months
  specifically assess the evolution of this parameter a few days before the occurrence of complications (occurrence of infection or graft rejection)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles JEBRAK, Doctor, Principal Investigator — Hôpital Bichat 75018 Paris
Locations (1):
- Jebrak, Paris, France